CLINICAL TRIAL: NCT04772209
Title: Comparison of Effectiveness and Complications of Heparin and Sodium Bicarbonate Catheter Lock Solutions in Non-Tunneled Hemodialysis Catheters
Brief Title: Comparison of Effectiveness and Complications of Catheter Lock Solutions in Non-tunneled Hemodialysis Catheters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zonguldak Ataturk State Hospital (Other)
Collaborators: Cumhuriyet University (Other); Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, mahmud islam, Medical Director of Nephrology clinic, Zonguldak Ataturk State Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ZADH-1
Record Dates: First submitted 2021-02-15; First posted 2021-02-26 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Catheter Blockage; Catheter-Related Infections; Dialysis Catheter; Thrombosis; Catheter Infection; Catheter Related Complication; Catheter Dysfunction
Keywords: catheter lock solution; sodium bicarbonate; heparin; Non-tunneled dialysis catheter
MeSH Terms: conditions — Catheter-Related Infections; Thrombosis | interventions — Sodium Bicarbonate; Heparin

STUDY DESIGN:
Intervention Model Description: Bicarbonate vs Heparin group (femoral vs jugular catheter)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sodium bicarbonate Arm (Active Comparator): In this arm, the catheter lock solution is sodium bicarbonate
  Interventions: Drug: Sodium bicarbonate
- Heparin arm (Active Comparator): In this arm, classic heparin will be used as a reference catheter lock solution (standard lock solution)
  Interventions: Drug: Heparin

INTERVENTIONS:
Drug: Sodium bicarbonate — Dialysis catheter lumen will be filled (locked) by sodium bicarbonate solution. The amount of solution depends on the diameter and length and will be in accordance with the manufacturer's specifications.
  Arms: Sodium bicarbonate Arm
Drug: Heparin — Dialysis catheter lumen will be filled (locked) by classic heparin. The amount of pure heparin depends on the diameter and length and will be in accordance with the manufacturer's specifications.
  Arms: Heparin arm

SUMMARY:
In our study, investigators will investigate the effectiveness and complications of two catheter lock solutions one of which is the standard heparin routinely used in comparison to Sodium bicarbonate. Both solutions were used but not compared head to head. Investigators aim to compare both solutions in terms of catheter lumen patency and their effect on catheter-related infections.

DETAILED DESCRIPTION:
The most important problem in patients with end-stage renal disease or patients with acute renal failure needing urgent hemodialysis treatment is the lack of appropriate vascular access. In acute situations, vascular access is usually provided by non-tunneled catheters. Main problems with this temporaray vascular access is failure due to lumen thrombosis. anther major problem is catheter related infection. In some patients, there is a handicap of using heparin. In some situations, heparin is not preferred for use. In terms of the probable shortage of resources and cost-effectiveness, Investigators aimed to compare head to head the superiority and non-inferiority of each solution. Sodium bicarbonate was compared to the isotonic solution and found to be effective for a short time. The main aim of this study is to compare both classic Heparin and sodium bicarbonate in Femoral and Jugular catheters aimed for dialysis. In both arms, the maximum patency and the observed side effects will be recorded. The maximal time used will be recorded. statistical analysis will be planned to compare the two groups.

ELIGIBILITY:
Inclusion Criteria:

* All patients over 18 years who assign consent will be included

Exclusion Criteria:

* patients less than 18 years of age
* Patients with active arterial or venous thrombosis problems
* Thrombocytopenic patients
* Patients with hypercoagulable states
* Patients with contraindications to heparin usage

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 441 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Time to first catheter failure (day) | 6 months
  The time from first sucessful dialysis session to the last one (in days)
Total Duration of catheter usage (day) | 6 months
  some patients need only 1-2 dialysis sessions while others may need too many sessions. In some cases a total of three dialysi sessions is whithin 3-4 days while others may need that number in wider range (e.g 10-14 days). Here both number and duraion effect is evaluated
Number of participants with catheter occlusion | 6 months
  The number of cases early catheter
Number of patients with catheter related infection | 6 months
  any catheter related infection(exit site, lumen inection etc) will be recorded
Time of catheter occlusion or failure | 6 months
  catheteres occluded by thrombi will be documented
Causes of premature catheter malfunction | 6 months
  any catheter needing exchange prematurly will be be evaluated for mulfunction cause (etiher mechanical thromus or kink rtc.)

SECONDARY OUTCOMES:
Total number of dialysis sessions with active patent catheter usage | 6 months
  In some cases intensive treatment is indicated. the effect of frequent usage of catheteres will be evaluated
Number of cases with venous thrombosis | 6 months
  catheters especially femoral have a risk of venous thrombosis, any clincal sign of thrombosis will be recorded. In case of catheter removal doppler ultrasound will be documented.

CONTACTS AND LOCATIONS:
Overall Officials: MAHMUD M ISLAM, MD, Principal Investigator — Zonguldak Ataturk State Hospital
Locations (2):
- Turkey (Türkiye) (2):
  - Cumhuriyet University Hospital, Sivas, TN
  - Zonguldak ataturk state hospital, Zonguldak, TN

IPD SHARING:
Plan to Share IPD: Yes
The study protocol and methods will be available in a paper intended for publication, any materials or data may be available on demand
Supporting Information: Study Protocol
Time Frame: Starting in February 2021 ends in September 2021
Access Criteria: The inquired information will be sent by e-mail

REFERENCES:
- [Background] El-Hennawy AS, Frolova E, Romney WA. Sodium bicarbonate catheter lock solution reduces hemodialysis catheter loss due to catheter-related thrombosis and blood stream infection: an open-label clinical trial. Nephrol Dial Transplant. 2019 Oct 1;34(10):1739-1745. doi: 10.1093/ndt/gfy388. PMID 30668833
- [Derived] Islam M. Sodium bicarbonate is a potential alternative to classic heparin as a lock solution for non-tunneled dialysis catheters: a result from the prospective randomized BicarbLock trial. Int Urol Nephrol. 2024 Apr;56(4):1465-1474. doi: 10.1007/s11255-023-03821-9. Epub 2023 Oct 12. PMID 37823971